CLINICAL TRIAL: NCT06025994
Title: Standardizing the Management of Patients with Coronary Microvascular Dysfunction: the SAMCRO Trial
Brief Title: Standardizing the Management of Patients with Coronary Microvascular Dysfunction
Acronym: SAMCRO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorzio Futuro in Ricerca (Other)
Collaborators: Università degli Studi di Ferrara (Other); Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 488/2023/Sper/AOUFe
Record Dates: First submitted 2023-08-15; First posted 2023-09-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Microvascular Angina; Microvascular Ischemia of Myocardium
Keywords: angina in non obstructive coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Microvascular Angina

STUDY DESIGN:
Intervention Model Description: The " Standardizing the Management of patients with Coronary Microvascular Dysfunction (SAMCRO) " trial is an all comers, prospective, randomized, multicenter, open-label study with blinded adjudicated evaluation of endpoints (PROBE).
Who Masked: Outcomes Assessor
Masking Description: The investigators in charge of follow-up visits and questionnaire collections will be different from investigators in charge of recruitment, baseline questionnaires collection and randomization procedure. The investigators in charge of follow-up procedures will be completely blinded to the randomization, as well as patient identifying information. Regarding clinical outcomes, an independent Clinical Event Committee (CEC) will adjudicate all endpoints. The CEC members and the CEC management team will be completely blinded to the randomization, as well as patient identifying information. Other measures to avoid or minimize bias introduced by the open-label design will include intent-to-treat principles of analysis and use of objective measures for endpoint classification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STANDARD OF CARE (No Intervention): Patients randomized to the control group will be managed according to current guidelines
- MULTI-DOMAIN LIFESTILE INTERVENTION (Experimental): Patients will receive five different kinds of intervention:
  i) strict management of CV and metabolic risk factors, ii) tailoring of medical therapy on the basis of the invasive assessment of CMD and coronary vasomotion, iii) dietary counselling, iv) exercise training v) psychological counselling
  Interventions: Other: MULTI-DOMAIN LIFESTILE INTERVENTION

INTERVENTIONS:
Other: MULTI-DOMAIN LIFESTILE INTERVENTION — All participants in the multi-domain lifestyle group will receive five different kinds of intervention: i) strict management of CV and metabolic risk factors, ii) tailoring of medical therapy on the basis of the invasive assessment of CMD and coronary vasomotion, iii) exercise training iv) dietary counselling, v) psychological intervention.
  Arms: MULTI-DOMAIN LIFESTILE INTERVENTION

SUMMARY:
The SAMCRO is an all comers, prospective, randomized, multicenter, open-label study with blinded adjudicated evaluation of outcomes (PROBE). The diagnosis of angina in non obstructive coronary artery disease (ANOCA) will be confirmed with coronary artery angiography and with the invasive assessment of coronary microvascular dysfunction (CMD) and coronary vasomotion. At least 120 ANOCA patients with invasively confirmed CMD will be randomized to i) multi-domain lifestyle intervention (experimental arm) vs. ii) standard of care (control arm). All patients will undergo follow-up visits at 6, 12, 24, 36, 48 and 60 months. The study endpoints will be the improvement of angina status and quality of life as assessed by validated questionnaires at one year. All participants in the multi-domain lifestyle group will receive five different kinds of intervention: i) dietary counselling, ii) strict management of cardiovascular (CV) and metabolic risk factors, iii) tailoring of medical therapy on the basis of the invasive assessment of CMD and coronary vasomotion, iv) exercise training and v) psychological intervention. Patients randomized to the control group will be managed according to current guidelines. The angina status will be assessed by the Seattle Angina Questionnaire (SAQ). Quality of life will be assessed using the EuroQoL (EQ5D-5L). Anxiety and depression will be assessed using the Beck Depression Inventory (BDI).

DETAILED DESCRIPTION:
The aim of the SAMCRO trial is to determine whether a multidomain lifestyle intervention improves angina status and quality of life in ANOCA patients as compared to current standard of care.

Patients will be randomized to:

EXPERIMENTAL ARM: MULTI-DOMAIN LIFESTILE INTERVENTION

Patients will receive five different kinds of intervention:

i) strict management of CV and metabolic risk factors, ii) tailoring of medical therapy on the basis of the invasive assessment of CMD and coronary vasomotion, iii) dietary counselling, iv) exercise training v) psychological counselling CONTROL ARM: STANDARD OF CARE Patients randomized to the control group will be managed according to current guidelines

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to hospital for chronic coronary syndrome (CCS) with indication for coronary artery angiography
* absence of obstructive coronary artery disease at invasive coronary artery angiography
* Coronary microvascular dysfunction as identified by invasive coronary physiology

Exclusion Criteria:

* Planned coronary revascularization
* Co-morbidity reducing life expectancy to less than 1 year
* Any factor precluding 1-year follow-up
* Prior Coronary Artery Bypass Graft (CABG) surgery
* Presence of a chronic total occlusion (CTO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2029-02-04 (Estimated)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire | 1-year
  The primary efficacy endpoint is the value of Seattle Angina Questionnaire (SAQ) summary score. The SAQ-SS ranges from 0 to 100 and higher values indicate better outcome

SECONDARY OUTCOMES:
EQ visual analogue scale | 1-year
  The continuous value of EQ visual analogue scale (EQ-VAS). The EQ-VAS scale ranges from 0 to 100 and higher values indicate better outcome
Beck Depression Inventory (BDI) | 1-year
  The continuous value of Beck Depression Inventory (BDI). BDI score ranges from 0 to 63. Higher scores indicate greater depressive severity.
Clinical adverse events | 1-year
  Cumulative occurrence of death, and hospital admission for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Campo, Principal Investigator — University Hospital of Ferrara
Locations (2):
- Italy (2):
  - AOU Ferrara, Ferrara, Ferrara
  - AOU di Parma, Parma, Parma

IPD SHARING:
Plan to Share IPD: Undecided